CLINICAL TRIAL: NCT01885780
Title: Phase IV Study_Prospective Evaluation of the Effectiveness of the Femtosecond Laser-assisted Refractive Astigmatic Keratotomy Following the Cataract Surgery.
Brief Title: Prospective Evaluation of the Effectiveness of the Femtosecond Laser-assisted Refractive Astigmatic Keratotomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1212
Record Dates: First submitted 2013-06-11; First posted 2013-06-25 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Astigmatism
Keywords: Astigmatism, arcuate incisions, astigmatic keratotomy
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Astigmatic keratotomy (Experimental)
  Interventions: Device: Laser-assisted Astigmatic keratotomy

INTERVENTIONS:
Device: Laser-assisted Astigmatic keratotomy — Laser-assisted Astigmatic keratotomy are performed by the VICTUS™ Femtosecond Laser Platform.

SUMMARY:
This clinical phase IV study is an open, prospective phase IV study and acts to evaluate the effectiveness of the femtolaser-assisted astigmatic keratotomy.

DETAILED DESCRIPTION:
The purpose of this prospective phase IV study acts to address the predictability and effectiveness of astigmatic keratotomy in eyes after femtolaser-assisted cataract surgery. Within this prospective data collection the laser-assisted Arcuate Incisions are performed by the VICTUS™ Femtosecond Laser Platform.

This study will be conducted at Gemini eye clinic in Zlin, Czech Republic by Dr. Pavel Stodulka who will treat up to 50 eyes. Patients will be recruited according to the study inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Clear corneal media
* Patients must be at least 40 years of age
* Mono- or bilateral Cataract treatment
* Keratometric astigmatism: ≥ 1.0 D and ≤ 3 D
* Patients must have read, understood the Patient Information and signed the informed consent form
* Patients are willing and able to return for follow-up examinations

Exclusion Criteria:

* The maximum K- value may not exceed 60D, the minimal value may not be smaller than 37D
* Pachymetry data for 7-8 mm zone are not available.
* Corneal disease or pathology, such as corneal scaring or opacity, that precludes transmission of laser wavelength or that distorts laser light
* Subjects with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally
* Lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Manifest Glaucoma
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye
* Known sensitivity to planned concomitant medications
* Patients regularly taking medicines that could influence the result of the treatment respectively the vision
* Patients with disorders of the ocular muscle, such as nystagmus or strabismus
* Patients with keratoconus, keratectasia or other irregular cornea changes
* Patients with connective tissue weakness
* Patients who are blind on one eye
* Subjects who are immune compromised or carrying diagnosis of connective tissue disease, clinically significant atopic disease, insulin dependent diabetes mellitus, autoimmune diseases, ocular herpes zoster or simplex, endocrine diseases, lupus, rheumatoid arthritis, collagenosis and other acute or chronic illnesses that will increase the risk to the subject or confound the outcomes of this study.
* Abnormal examination results from slit lamp, fundus examination or IOL Master, age related changes are acceptable
* Patients with eye diseases which decreases the visual acuity such as macular degeneration, macular edema, proliferative diabetic Retinopathy
* Abnormal examination results from Topography, age related changes are acceptable
* Patients who are pregnant or nursing
* Patients with concentration disorders, epilepsy and other complicating diseases
* Patients who are participating in another clinical study 30 days before

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Keratomic corneal astigmatism | The study endpoints will be calculated for the 3-Months follow-up examination.
  The postoperative keratomic corneal astigmatism is in 60% of all eyes equal or better than 1.0D

SECONDARY OUTCOMES:
Topographic corneal and subjective cylinder | This end point is measured at the 3 Months Follow Up.
  * The postoperative astigmatism in topography is in 60% of all eyes equal or better than 1.0D
  * The postoperative subjective astigmatism in manifest refraction is in 60% of all eyes equal or better than 1D.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodulka, Dr. med, Principal Investigator — Gemini clinic, Zlin; Pavel Stodulka, Dr. med, Principal Investigator — Gemini Eye Clinic
Locations (1):
- Gemini Eye Clinic, Zlín, Czechia